CLINICAL TRIAL: NCT04743479
Title: Artificial Intelligence-based Health Information Management System and Key Technology Study of Early Screening and Hierarchical Diagnosis and Treatment of Pancreatic Cancer
Brief Title: Artificial Intelligence-based Early Screening of Pancreatic Cancer and High Risk Tracing (ESPRIT-AI)
Acronym: ESPRIT-AI
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Associated Professor at the Institute of Pancreatic Surgery, Changhai Hospital
Other Study IDs: ChanghaiH-PP07
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer; Diabetes; Familial Pancreatic Cancer; Pancreatic Cystic Neoplasm; Chronic Pancreatitis; Hereditary Pancreatitis
Keywords: Screening; Early Diagnosis; Artificial Intelligence; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Diabetes Mellitus; Pancreatic carcinoma, familial; Pancreatitis, Chronic; Hereditary pancreatitis; Disease | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients in this study will have the option of donating blood for biobanking, approximately 10cc of plasma and 10cc of serum. Further, samples that are routinely collected for diagnostic purposes may be collected and banked at the time of their clinically routine procedure. If a patient consents to the use of extra material for research purposes, the biological samples will be banked and the blood, and/or pancreatic juice/cystic fluid, tissues, and saliva will be used for identification and characterization of potential biomarkers from de-identified samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- New Onset Diabetes: New Onset Diabetes must meet one of the following criteria:
  1. Documented diabetes diagnosed within the past 3 years.
  2. Definite new-onset diabetes based on recent fasting blood glucose (FBG) values ≥126 mg/dl (7.0 mmol/L) or Hemoglobin A1c (HbA1c) ≥ 6.5%. All glycemic parameters must be measured in an outpatient setting.
  Interventions: Diagnostic Test: high-resolution MRI/CT examinations
- Familial pancreatic cancer: Familial pancreatic cancer must meet one of the following criteria:
  1. ≥ 2 blood relatives with pancreatic cancer (includes 1st-3rd degree relatives)
  2. One 1st degree relative with PDAC diagnosed before age 60
  Interventions: Diagnostic Test: high-resolution MRI/CT examinations
- Inherited syndromes associated with pancreatic cancer: Family history includes with inherited syndromes associated with pancreatic cancer ( ≥ 2 blood relative, includes 1st-3rd degree relatives).
  Inherited syndromes must meet one of the following criteria:
  1. Hereditary pancreatitis
  2. Familial atypical multiple mole and melanoma syndrome
  3. Hereditary nonpolyposis colon cancer
  4. Peutz-Jeghers syndrome
  5. Hereditary breast and ovarian cancer syndromes
  Interventions: Diagnostic Test: high-resolution MRI/CT examinations
- Pancreatic Cystic Neoplasm: Pancreatic Cystic Neoplasm, including intraductal papillary mucinous neoplasms (IPMN) and mucinous cystic neoplasms (MCN), which are defined by endoscopic ultrasound or serial imaging.
  Interventions: Diagnostic Test: high-resolution MRI/CT examinations
- Chronic pancreatitis: Chronic pancreatitis, defined by cross-sectional imaging, endoscopic ultrasound, functional testing abnormalities OR as diagnosed by a gastroenterologist.
  Interventions: Diagnostic Test: high-resolution MRI/CT examinations

INTERVENTIONS:
Diagnostic Test: high-resolution MRI/CT examinations — Participants will undergo annual questionnaire survey, laboratory tests and high-resolution MRI/CT examinations of the pancreas. Any suspicious lesions will be further examined by endoscopic ultrasound (EUS).
  Other Names: questionnaire survey; laboratory tests

SUMMARY:
Pancreatic cancer is one of the most fatal malignancies with a 5-year survival rate of only ~6%[1]. The reasons for this high mortality rate can be attributed to several factors, of which perhaps the most important is delayed diagnosis due to vague symptoms and consequently missed opportunities for surgical resection. Therefore, the ability to detect pancreatic cancer at an early, more curable stage is urgently needed.

Identifying risk factors and biomarkers of early pancreatic cancer could facilitate screening for individuals at higher than average risk and expedite the diagnosis in individuals with symptoms and substantially improve an individual's chance of surviving the disease. Thus, the investigators propose this longitudinal study entitled, "Artificial Intelligence-based Early Screening of Pancreatic Cancer and High Risk Tracing (ESPRIT-AI)" in order to generate clinical data sets and bank serial blood specimens of high risk individuals.

DETAILED DESCRIPTION:
The study is being run by a team of dedicated physicians and researchers, led by Jin Gang, MD, Director of Department of general surgery of Shanghai Changhai Hospital. The trial will include individuals with new-onset diabetes (diagnosed within the past 3 year), familial pancreatic cancer, inherited syndromes associated with pancreatic cancer (including hereditary pancreatitis, familial atypical multiple mole and melanoma syndrome, hereditary nonpolyposis colon cancer, Peutz-Jeghers syndrome, hereditary breast and ovarian cancer syndromes, etc), pancreatic cystic neoplasm (including IPMN, MCN) as well as chronic pancreatitis. Participants will undergo annual laboratory tests and high-resolution MRI/CT examinations of the pancreas. Any suspicious lesions will be further examined by endoscopic ultrasound (EUS). If pancreatic cancer or a pre-cancerous lesion is identified, the individual will be referred for surgery. We will also be collecting a blood sample from all participants for DNA isolation. Clinical data and biological specimens contained in this study may be used for a wide variety of future related studies to the cause, diagnosis, outcome and treatment of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to provide informed consent and sign an informed consent form.
* Subject or authorized representative must be willing to complete a detailed questionnaire.
* Subject must meet one of the following criteria:

  1. New onset diabetes (diagnosed within the past 3 years)
  2. Familial pancreatic cancer
  3. Inherited syndromes associated with pancreatic cancer (including Hereditary pancreatitis, Familial atypical multiple mole and melanoma syndrome, Hereditary nonpolyposis colon cancer, Peutz-Jeghers syndrome, Hereditary breast and ovarian cancer syndromes, etc)
  4. Pancreatic cystic neoplasm (including IPMN, MCN)
  5. Chronic pancreatitis

Exclusion Criteria:

* Subject has been diagnosed with pancreatic cancer or other malignant tumors in the last 5 years;
* Subject has any medical condition that contraindicates high-resolution MRI or CT;
* Subject cannot be followed up or is participating in other clinical trials.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High risk individuals of pancreatic cancer
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence | 5 years
  Determine incidence of pancreatic cancer or precursor lesions among high risk individuals.
Hazard ratio (HR) | 5 years
  Assesses the influence of risk factors on the incidence of pancreatic cancer or precursor lesions among high risk individuals.

SECONDARY OUTCOMES:
Survival time | 5 years
  Calculate survival time from point of diagnosis and treatment among the identified patients with pancreatic cancer.
HR | 5 years
  Assesses the influence of risk factors on survival time among the identified patients with pancreatic cancer.
Diagnostic yield | 5 years
  Determine diagnostic yield (sensitivity, specificity, positive/negative predictive value and accuracy) of AI-based surveillance program to predict early stage pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, M.D., Study Chair — Department of general surgery, Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamisawa T, Wood LD, Itoi T, Takaori K. Pancreatic cancer. Lancet. 2016 Jul 2;388(10039):73-85. doi: 10.1016/S0140-6736(16)00141-0. Epub 2016 Jan 30. PMID 26830752
- [Background] Lin QJ, Yang F, Jin C, Fu DL. Current status and progress of pancreatic cancer in China. World J Gastroenterol. 2015 Jul 14;21(26):7988-8003. doi: 10.3748/wjg.v21.i26.7988. PMID 26185370
- [Background] Henrikson NB, Aiello Bowles EJ, Blasi PR, Morrison CC, Nguyen M, Pillarisetty VG, Lin JS. Screening for Pancreatic Cancer: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2019 Aug 6;322(5):445-454. doi: 10.1001/jama.2019.6190. PMID 31386140
- [Background] Singhi AD, Koay EJ, Chari ST, Maitra A. Early Detection of Pancreatic Cancer: Opportunities and Challenges. Gastroenterology. 2019 May;156(7):2024-2040. doi: 10.1053/j.gastro.2019.01.259. Epub 2019 Feb 2. PMID 30721664
- [Background] Pereira SP, Oldfield L, Ney A, Hart PA, Keane MG, Pandol SJ, Li D, Greenhalf W, Jeon CY, Koay EJ, Almario CV, Halloran C, Lennon AM, Costello E. Early detection of pancreatic cancer. Lancet Gastroenterol Hepatol. 2020 Jul;5(7):698-710. doi: 10.1016/S2468-1253(19)30416-9. Epub 2020 Mar 2. PMID 32135127
- [Background] Maitra A, Sharma A, Brand RE, Van Den Eeden SK, Fisher WE, Hart PA, Hughes SJ, Mather KJ, Pandol SJ, Park WG, Feng Z, Serrano J, Rinaudo JAS, Srivastava S, Chari ST; Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC). A Prospective Study to Establish a New-Onset Diabetes Cohort: From the Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer. Pancreas. 2018 Nov/Dec;47(10):1244-1248. doi: 10.1097/MPA.0000000000001169. PMID 30325864